CLINICAL TRIAL: NCT06198634
Title: Post Intubation Laryngeal Hazards in Children in the Pediatric Intensive Care Unit
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ashrakt Ahmed Mahmoud, principal investigator, Assiut University
Other Study IDs: intubation laryngeal hazard
Record Dates: First submitted 2023-12-23; First posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-12

CONDITIONS: Laryngeal Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
this study aims to detect the effect of endotracheal intubation on the larynx of the pediatric population in order to allow early detection of any hazards

DETAILED DESCRIPTION:
Laryngeal lesions in children can be caused by a number of risk factors, including patient variables (prematurity, cardiac comorbidities), intubation method (in an emergency, by an unskilled team), and endotracheal tube use. (large size, cuffed tube), longer duration of intubation, infection, and insufficient patient sedation are just a few risk factors that can contribute to the development of laryngeal lesions in children. Endoscopic imaging of the larynx is essential in pediatric intubation-related laryngeal injuries since the intensity of symptoms may not necessarily be correlated with the extent of laryngeal injury that is actually present. Therefore, after intubation, we will evaluate neonates, babies, and kids who have laryngeal problems. The flexible fiberoptic nasopharyngo-laryngoscope, or laryngoscopy, is the preferred technique to assess these children's issues and represents a substantial development in the diagnosis of laryngeal pathology in children. As well as rigid bronchoscopy and direct laryngoscopy, under general anesthesia. The risks associated with anesthesia and instrumentation are two key drawbacks of this method. Without transferring to the operating room or requiring general anesthesia, the infant can be assessed in the outpatient clinic. Direct observation of the nasopharynx and larynx in a professional environment

ELIGIBILITY:
Inclusion Criteria:

1. Age: from 2 month to 18 year
2. Gender: both sexes will be included in the study
3. Endotracheal intubation in emergency or elective sitting for 24hr or more

Exclusion Criteria:

* 1-Congenital laryngeal lesions 2-Head and neck surgery 3-CNS infections 4-Craniofacial malformations

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: the patients will the pediatric population who underwent endotracheal intubation in emergency or elective sitting for 24hr or more
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-01-15 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
measurement of pediatric post intubation laryngeal lesions | 7_10 days post_intubation
  measurement of presence or absence of laryngeal lesions (supraglottic,glottic,subglottic) post intubation in pediatrics using fiberoptic naso_pharyngeal_laryngoscopy

REFERENCES:
- [Background] Lambercy K, Pincet L, Sandu K. Intubation Related Laryngeal Injuries in Pediatric Population. Front Pediatr. 2021 Feb 10;9:594832. doi: 10.3389/fped.2021.594832. eCollection 2021. PMID 33643969
- [Background] Lindholm CE. Prolonged endotracheal intubation. Acta Anaesthesiol Scand Suppl. 1970;33:1-131. doi: 10.1111/j.1399-6576.1969.tb00750.x. No abstract available. PMID 5459079
- [Background] Veder LL, Joosten KFM, Schlink K, Timmerman MK, Hoeve LJ, van der Schroeff MP, Pullens B. Post-extubation stridor after prolonged intubation in the pediatric intensive care unit (PICU): a prospective observational cohort study. Eur Arch Otorhinolaryngol. 2020 Jun;277(6):1725-1731. doi: 10.1007/s00405-020-05877-0. Epub 2020 Mar 4. PMID 32130509